CLINICAL TRIAL: NCT06682039
Title: Anxiety and Negative Attentional Bias in Adolescent and Young Adult Cancer Survivors
Brief Title: Attention Bias Modification for the Improvement of Anxiety in Adolescent and Young Adult Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RG1124389; NCI-2024-06745 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA015704 (NIH); STUDY00004811 (Other: Fred Hutch/University of Washington/Seattle Children's Cancer Consortium)
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Childhood Hematopoietic and Lymphatic System Neoplasm; Childhood Malignant Solid Neoplasm
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blind to study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (ABM) (Experimental): Patients engage in ABM over 10 minutes BIW and respond daily to text messaging prompts for 4 weeks.
  Interventions: Other: Internet-Based Intervention; Other: Interview; Other: Questionnaire Administration; Other: Text Message-Based Navigation Intervention
- Arm II (inert attention task) (Active Comparator): Patients engage in inert attention task sessions over 10 minutes BIW for 4 weeks. Patients also receive and respond to text messaging prompts QD for 4 weeks. After completion of the 4 week follow up survey, patients are given access to all components of ABM and texts on study.
  Interventions: Other: Internet-Based Intervention; Other: Questionnaire Administration; Other: Text Message-Based Navigation Intervention

INTERVENTIONS:
Other: Internet-Based Intervention — Engage in ABM + text messaging prompts
  Arms: Arm I (ABM)
Other: Internet-Based Intervention — Engage in inert attention task sessions
  Arms: Arm II (inert attention task)
Other: Interview — Ancillary studies
  Arms: Arm I (ABM)
Other: Questionnaire Administration — Ancillary studies
Other: Text Message-Based Navigation Intervention — Participants will respond to daily messaging prompts.
  Other Names: Automated Text Message-Based Navigation; Text Message-Based Navigation

SUMMARY:
This clinical trial studies how well attention bias modification (ABM) improves anxiety in adolescent and young adult (AYA) cancer survivors. Cancer-related anxiety is the most prevalent mental health problem affecting AYA cancer survivors. Cancer-related anxiety is associated with long-term negative outcomes such as poor quality of life, depression, distress, substance use, sleep problems, fatigue, and pain. ABM uses techniques to help patients change the way they react to environmental triggers that may cause a negative reaction. ABM uses brief self-guided smartphone applications. Patients complete repetitive association reaction-time tasks targeting automatic and unconscious negative attention biases to retrain attention away from perceived threat and towards a neutral or positive stimuli. Gratitude-finding and savoring activities are also provided to maintain and increase positive emotions. Using ABM plus gratitude-finding and savoring activities may improve anxiety in AYA cancer survivors.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients engage in ABM over 10 minutes twice a week (BIW) and respond daily to text messaging prompts activity for 4 weeks.

ARM II: Patients engage in inert attention task sessions over 10 minutes BIW for 4 weeks. Patients also receive and respond to text messaging prompts QD for 4 weeks.

After completion of study intervention, patients are followed up at 4 weeks. After completion of this 4 week follow up survey, patients are given access to all components of ABM and texts on study.

ELIGIBILITY:
Inclusion Criteria:

* Age 15-29 years
* Diagnosis of cancer malignancy
* Received active/curative cancer treatment OR received/actively receiving cancer survivorship care at Seattle Children's Hospital (SCH) or other study referring site (e.g. St. Jude)
* Currently off active/curative cancer treatment
* Patient able to understand/read/write English language
* Cognitively able to participate in ABM intervention and complete surveys
* Patient has access to smartphone able to send and receive text messages
* Patient has access to computer or smartphone for Inquisit program

Exclusion Criteria:

* Patients on active/curative cancer treatment
* Cognitively or physically unable to participate in ABM intervention and surveys
* Patients who cannot understand/read/write English will be excluded from the research because the ABM intervention is currently only available in English
* Furthermore, patients who do not have access to technology (smartphone/computer) will be excluded from the study as this technology is absolutely required to engage in the study intervention

Ages: 15 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2024-11-08 (Actual); Primary Completion 2026-01-12 (Actual); Study Completion 2026-01-12 (Actual)

PRIMARY OUTCOMES:
Clinic recruitment rates | Up to 4 weeks post-intervention
  Feasibility will be assessed via clinic recruitment rates, defined as (number [#] of adolescent and young adults [AYAs] who enroll in the study) / (total # of AYAs screened as eligible). Attention bias modification (ABM) will be considered feasible with ≥ 50% enrollment.
Retention rates | Up to 4 weeks post-intervention
  Uptake will be assessed via retention rates, defined as (# of AYAs who complete 4-week treatment duration of ABM) / (# of AYAs who enroll in the study). ABM will be considered feasible with ≥ 70% retention.
Patient acceptability of ABM: Client Satisfaction Questionnaire (CSQ-8) | At 4 weeks post intervention
  Will be assessed using the Client Satisfaction Questionnaire (CSQ-8). The CSQ-8 is an 8-item questionnaire used to assess level of satisfaction with care. Items are scored on a Likert scale from 1 (low satisfaction) to 4 (high satisfaction) with different descriptors for each response point. Total scores range from 8 to 32, with higher scores indicating greater satisfaction(scores ≥26 indicate satisfaction).
Patient acceptability of ABM: System Usability Scale (SUS) | At 4 weeks post intervention
  Will be assessed using the System Usability Scale (SUS). The SUS is a well-validated and widely used 10-item scale to evaluate the perceived usability of digital interventions. Items are rated on a 5-point Likert scale for a total score ranging from 0-100, and scores ≥ 70 considered adequate usability.

OTHER OUTCOMES:
Change in Health-Related Quality of Life from Baseline to Post-treatment as Assessed by PROMIS Profile-57 | From baseline to post-treatment (4 weeks)
  PROMIS Profile-57: The Patient-Reported Outcomes Measurement Information System (PROMIS) are publicly available, rigorously tested, and well-validated measures supported by the NIH Common Fund. The PROMIS Profile-57 is a self-report measure covering the domains of physical function, anxiety, depression, fatigue, sleep disturbance, social participation, pain interference, and pain intensity.
Change in Resilience from Baseline to Post-treatment as Assessed by CD-RISC-10 | From baseline to post-treatment (4 weeks)
  Connor-Davidson 10 Resilience Scale (CD-RISC-10): The CD-RISC is a well-validated and widely used instrument to measure inherent resiliency. Questions revolve around personal problem-solving and approaches to adversity. The 10-item instrument has high internal consistency (Cronbach's alpha = 0.85), and has been used in diverse populations including adolescents, parents, and cancer patients. Each item consists of a 5-point Likert scale (scored from zero to four) for a total of 40 points, with higher scores reflecting greater resilience.
Change in Psychological Distress from Baseline to Post-treatment as Assessed by Kessler-6 | From baseline to post-treatment (4 weeks)
  Kessler-6 Psychological Distress Scale (K6): This 6-item scale measures "level of psychological distress experienced in the past month." It was developed for the US National Health Interview Survey, and is currently being used in Canada, Australia and world-wide as part of the World Health Organization (WHO) world mental health initiative. The instrument strongly discriminates between community cases and non-cases of Diagnostic and Statistical Manual of Mental Disorder (DSM)-V psychiatric disorders such as serious emotional distress or serious mental illness. It has been extensively cross-validated, including among adolescents. Responses are scored on a 5-point Likert scale, generating a range of zero to 24 points. Previous studies have shown that scores ≥ 7 are consistent with "high" distress and those ≥ 13 meet criteria for serious, or debilitating psychological distress.
Change in Anxiety and Depression Symptoms from Baseline to Post-treatment as Assessed by HADS-6 | From baseline to post-treatment (4 weeks)
  Hospital Anxiety and Depression Scale (HADS): 14 items assess symptoms of anxiety and depression, respectively, in patients with serious illness. It has been validated in AYAs with chronic illness and cancer survivors, with excellent reliability (α=0.83-0.82). Items are scored 0-3 (subscale range 0-21), with scores ≥8 categorized as borderline abnormal, and ≥11 categorized as abnormal.
Change in Health Anxiety from Baseline to Post-treatment as Assessed by SHAI | From baseline to post-treatment (4 weeks)
  Short Health Anxiety Inventory (SHAI): The SHAI contains 14 items that assess health anxiety independent of physical health status. Items assess worry about one's health, awareness of bodily sensations and/or changes, and the feared consequences of having an illness. It can be used in both healthy individuals and physically ill individuals including those who were temporarily sick or diagnosed with a serious and/or chronic illness. The scale has been validated in clinical and non-clinical samples. Total score ranges from 0 to 42, with higher scores indicating greater health anxiety.
Change in Fear of Cancer Recurrence from Baseline to Post-treatment as Assessed by FCRI-SF | From baseline to post-treatment (4 weeks)
  Fear of Cancer Recurrence Inventory-SF (FCRI-SF): The FCRI-SF is a widely utilized and validated 9-item measure that evaluates the presence and severity of intrusive thoughts associated with fear of cancer recurrence. Each item is rated on a Likert scale ranging from 0 ("not at all" or "never") to 4 ("a great deal' or "all the time"). A higher score indicates higher levels of fear of cancer recurrence.
Change in Experience of Attention Bias from Baseline to Post-treatment as Assessed by ABQ | From baseline to post-treatment (4 weeks)
  The Attention Bias Questionnaire (ABQ) consists of nine items reflecting the subjective experience of attention bias towards threats, with two sub-scales: Engagement with Threat and Difficulty to Disengage from Threat. High ABQ scores are correlated with trait anxiety, social anxiety, PTSD, and depression. It has been validated in ages 18+, with high internal consistency (Cronbach's alpha=0.90). Total score ranges from 0 to 4, with higher scores indicating greater attention bias.
Change in Pain Intensity from Baseline to Post-treatment as Assessed by PROMIS Pain Intensity | From baseline to post-treatment (4 weeks)
  PROMIS Pain Intensity: The Patient-Reported Outcomes Measurement Information System (PROMIS) are publicly available, rigorously tested, and well-validated measures supported by the NIH Common Fund. The PROMIS Pain Intensity (3-item) instrument assesses how much a person hurts.
Change in Pain Frequency, Intensity, and Interference from Baseline to Post-treatment | From baseline to post-treatment (4 weeks)
  3 questions will assess pain frequency (6- or 7-item Likert scale from "not at all" to "daily"), pain intensity (11-point NRS, 0-10), and pain interference (11-point NRS, 0-10).
Change in Pain-related Activity Limitations from Baseline to Post-treatment as Assessed by CALI-9 | From baseline to post-treatment (4 weeks)
  Child Activity Limitations Interview-9 (CALI-9): The CALI-9 is a brief measure for assessing activity limitations in children and adolescents with chronic pain. This measure has demonstrated good internal consistency and high cross-informant reliability. Total score ranges from 0-100, with higher scores indicating greater pain-related activity limitations.
Change in Overall Sleep Quality Score from Baseline to Post-treatment as Assessed by ASWS-SF | From baseline to post-treatment (4 weeks)
  The Adolescent Sleep Wake Scale Short Form (ASWS-SF) is a 10-item measure of behavioral sleep patterns that has been validated in general adolescent populations. The measure provides an overall sleep quality score, and 3 subscale scores: going to bed, falling asleep and reinitiating sleep, and returning to wakefulness. Items are rated on a 6-point Likert scale, and averaged to compute subscale and total measure scores. Total scores range from 1 to 6 with higher scores indicating better sleep quality.
Change in Insomnia Symptoms from Baseline to Post-treatment as Assessed by AIQ | From baseline to post-treatment (4 weeks)
  The Adolescent Insomnia Questionnaire (AIQ) is a 13-item screening measure of insomnia in adolescents. The measure has demonstrated strong reliability and high internal inconsistency. Items are rated on a 5-point Likert scale. Total scores range from 0 to 52 with higher scores indicating more insomnia symptoms.
Cognitive Function from Baseline to Post-treatment as Assessed by PROMIS NeuroQOL | Baseline
  PROMIS NeuroQOL Cognitive Function-SF: The Patient-Reported Outcomes Measurement Information System (PROMIS) are publicly available, rigorously tested, and well-validated measures supported by the NIH Common Fund. The PROMIS NeuroQOL Cognitive Function-SF measures perceived difficulties in everyday cognitive abilities such as memory, attention, and decision-making.
Change in Attention Bias Scores from Baseline to Post-treatment as Assessed by Dot Probe Task | From baseline to post-treatment (4 weeks)
  The Dot Probe Task is a well-established and widely utilized digitized reaction time test to measure attention bias towards threat. Attention bias scores will be computed by subtracting the mean reaction time in trials where probes replace negative stimuli from the mean reaction time in trials where probes replace neutral/positive stimuli. Positive attention bias scores will indicate an attentional bias towards threatening stimuli, and negative scores will indicate an attentional bias towards non-threatening stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lau, PhD, Principal Investigator — Fred Hutch/University of Washington/Seattle Children's Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington/Seattle Children's Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-09-19): https://cdn.clinicaltrials.gov/large-docs/39/NCT06682039/ICF_000.pdf